CLINICAL TRIAL: NCT01596010
Title: Single Dose, Double-blind, Two-way Cross-over Bioequivalence Trial With 2 Different Oral Formulations of Estradiol and Norethisterone
Brief Title: Investigation of 2 Different Oral Formulations of Estradiol and Norethisterone in Healthy Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KLI-1915; 2007-003350-28 (EudraCT Number)
Record Dates: First submitted 2012-05-09; First posted 2012-05-10 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Menopause; Healthy
MeSH Terms: interventions — Estradiol; Norethindrone Acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- New formulation (Experimental)
  Interventions: Drug: 2 mg estradiol / 1 mg norethisterone acetate (NETA)
- Old formulation (Active Comparator)
  Interventions: Drug: 2 mg estradiol / 1 mg norethisterone acetate (NETA)

INTERVENTIONS:
Drug: 2 mg estradiol / 1 mg norethisterone acetate (NETA) — A single dose of one tablet under fasting conditions separated by a wash-out period of 2 weeks (+0-2 days) between dosing visits. Administered orally.

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate whether a reformulated estradiol/norethisterone acetate (NETA) formulation is bioequivalent to that of Kliogest® (estradiol/norethisterone acetate (NETA) in healthy women.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal defined as at least 12 months spontaneous amenorrhoea, with serum FSH (follicle stimulating hormone) levels at least 40 IU/L and estradiol maximum 25 pg/mL. If the date of spontaneous amenorrhoea can not be identified because of previous hormone replacement therapy, serum FSH at least 40 IU/L and estradiol maximum 25 pg/mL
* Non-smoking
* Body Mass Index (BMI) maximum 35.0 kg/m^2
* Able to understand, read and speak German fluently
* Good state of health evidenced by medical history, physical examination including gynecological examination, and results from laboratory examination
* Willing to abstain from intake of caffeine containing food and beverages within 48 hours before drug administration

Exclusion Criteria:

* Known or suspected allergy to trial products or related products
* Previous use of oral, transdermal, nasal spray, vaginal preparations and implants within 8 weeks prior to the planned first drug administration
* Known, suspected or history of breast cancer
* Known or suspected estrogen dependent neoplasia e.g. endometrial cancer
* Abnormal genital bleeding of unknown aetiology
* Known insulin dependent as well as non-insulin dependent diabetes mellitus
* Positive test for HIV (human immunodeficiency virus) and/or hepatitis B and C
* Systolic blood pressure (BP) above or equal to 160 mm Hg and/or diastolic BP above or equal to 100 mm Hg, currently treated or untreated

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-10; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Area under the Curve (0-t) | Up to 72 hours after trial product administration
Cmax, maximum concentration | Up to 72 hours after trial product administration

SECONDARY OUTCOMES:
Time to maximum (tmax) | Up to 72 hours after trial product administration
Area under the curve from time zero to infinity | Up to 72 hours after trial product administration
Terminal half-life (t½) | Up to 72 hours after trial product administration
Terminal rate constant | Up to 72 hours after trial product administration
Incidence of adverse events (AEs) | Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Neu-Ulm, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com